CLINICAL TRIAL: NCT02580812
Title: Multicentric Observational National Analysis of Listeriosis and Listeria : Evaluation of the Neurological Consequences of Perinatal Listeriosis Infection
Brief Title: Neurological Consequences of Perinatal Listeriosis Infection
Acronym: MONALISABABY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P140940
Record Dates: First submitted 2015-08-31; First posted 2015-10-20 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Perinatal Listeriosis
Keywords: Perinatal listeriosis; Neurological impairment; Sepsis; Prematurity; Neurotropism; Listeria monocytogenes; Intellectual Quotient
MeSH Terms: conditions — Neurologic Manifestations; Sepsis; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MONALISA 5-years old children (Experimental): Clinical and neuropsychological evaluation procedure 90 children
  Interventions: Other: Clinical and neuropsychological evaluation procedure
- EPIPAGE 5 -years old children (Active Comparator): Cohort of prematurely borne children and their controls Clinical and neuropsychological evaluation procedure 270 children
  Interventions: Other: Clinical and neuropsychological evaluation procedure

INTERVENTIONS:
Other: Clinical and neuropsychological evaluation procedure — WPPSI, NEPSY, Brief, SDQ, Vineland and SCQ evaluation Clinical examination

SUMMARY:
The purpose of the study is to determine whether perinatal listeriosis is associated with long-term neurological consequences, and to evaluate the respective contribution of perinatal sepsis, of prematurity and of the known neurological tropism of the involved pathogen, Listeria monocytogenes.

DETAILED DESCRIPTION:
Perinatal listeriosis is defined by the occurrence of maternal listeriosis at birth and/or of early-onset listeriosis in the neonate (defined by the positive culture of any sample of maternal or neonatal origin).

Neurological involvement is defined by the presence of inflammation of the cerebrospinal fluid of positive culture or the cerebro-spinal fluid.

Evaluation is performed at the age of 5 years, and includes WPPSI evaluation of the Intelligence Quotient (IQ), NEPSY evaluation of the executive functions and clinical evaluation checking for any motor, sensorial or other focal deficiency among 90 cases and 270 controls matched for gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Children from the MONALISA cohort (culture proven-maternal listeriosis)
* Or Children from the EPIPAGE cohort (control group)
* Written consent from the parent(s) or legal representative

Exclusion Criteria:

* Children whose parents or legal representative would deny their consent

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Reduction of > 20 points of the Intellectual Quotient | Day 1
  Evaluated by standard tests (WPPSI-IV)

SECONDARY OUTCOMES:
Score obtained at M-ABC evaluation test (Movement-ABC) | Day 1
  to evaluate alteration of executive functions
Score obtained at SDQ evaluation test (Strenghts and Difficulties Questionnaire) | Day 1
  to evaluate alteration of cognitive functions
Score obtained at SCQ evaluation test (Social Communication Questionnaire) | Day 1
  to evaluate alteration of cognitive functions
Score obtained at BRIEF-P evaluation test (Behavior Rating Inventoring Executive Function) | Day 1
  to evaluate alteration of executive functions
Score obtained at HOME evaluation test (Home Observation and Measurement of Environment) | Day 1
Score obtained at Vineland Scale | Day 1
Scores obtained at NEPSY-2 evaluation tests | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Caroline CHARLIER-WOERTHER, MD, PhD, Principal Investigator — Service des Maladies Infectieuses et Tropicales, Centre d'Infectiologie Necker-Pasteur, IHU Imagine - Hôpital Necker-Enfants Malades, APHP / Centre National de Référence Listeria, Centre collaborateur OMS Listeria, Institut Pasteur; Marc LECUIT, MD, PhD, Study Chair — Service des Maladies Infectieuses et Tropicales, Centre d'Infectiologie Necker-Pasteur, IHU Imagine - Hôpital Necker-Enfants Malades, APHP /Centre National de Référence Listeria, Centre collaborateur OMS Listeria, institut Pasteur
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

REFERENCES:
- [Background] Charlier C, Barrault Z, Rousseau J, Kermorvant-Duchemin E, Meyzer C, Semeraro M, Fall M, Coulpier G, Leclercq A, Charles MA, Ancel PY, Lecuit M. Long-term neurological and neurodevelopmental outcome of neonatal listeriosis in France: a prospective, matched, observational cohort study. Lancet Child Adolesc Health. 2023 Dec;7(12):875-885. doi: 10.1016/S2352-4642(23)00195-5. Epub 2023 Oct 20. PMID 37871603